CLINICAL TRIAL: NCT05833516
Title: Operator Radiation Exposure in Hyper Adduction of Right Radial Artery/Arm vs Left Arm Drag Over Technique.
Brief Title: Hyper Adduction of Right Radial Artery/Arm vs Left Drag Over Technique
Acronym: HARRA
Status: Completed | Type: Observational
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: #2022-05-19
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Radiation Exposure
Keywords: prospective; randomized; radiation dose; operator exposure; cardiac catheterization
MeSH Terms: interventions — Cardiac Catheterization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hyperadducted Right Radial Arm (HARRA): The primary operators will wear real time radiation dose monitoring at the left eye, right eye, thorax and abdomen level. At the end of each diagnostic procedure the cumulative radiation dose (measured in µSv) data at each level will be collected. The radiation dose exposure in patients randomized to hyperadducted right radial arm will be recorded for primary outcome.
  Interventions: Diagnostic Test: Cardiac Catheterization
- Left Arm Drag over technique: The primary operators will wear real time radiation dose monitoring at the left eye, right eye, thorax and abdomen level. At the end of each diagnostic procedure the cumulative radiation dose (measured in µSv) data at each level will be collected. The radiation dose exposure in patients randomized to Left Arm drag over technique will be recorded for primary outcome.
  Interventions: Diagnostic Test: Cardiac Catheterization

INTERVENTIONS:
Diagnostic Test: Cardiac Catheterization — The cardiac catheterization is an invasive procedure in which right or left radial artery of patient will be accessed to obtain cardiac angiogram. The study participants are both operators and patients by obtaining the amount of radiation they both were exposed in these two different arm techniques.
  The patient will have to do nothing more than following the existing standard protocols which are followed nationwide. As, the radiation exposure to patients are already measured in the software itself. The operators however would be wearing radiation badges in 4 different anatomic locations to record radiation data for study.

SUMMARY:
Several studies have shown that operator exposure via left transradial catheterization has yielded less operator exposure compared to standard right transradial procedure. However, in light of new data, the investigators hypothesize a hyperadducted right arm during right transradial cardiac catheterization will yield comparable, or the same operator radiation exposure.

DETAILED DESCRIPTION:
Few studies have examined operator's radiation exposure tor transradial cardiac catheterization between the left vs right radial artery approach. In light of recent studies (Schiabasi et al) demonstrating adduction of the right arm yields lower operator exposure than that of the right arm positioned away from the body to the operators. The investigators seek to examine if hyper adduction of the right arm yields similar operator exposure to that of the left radial approach.

Historically the left radial approach has been more favorable in terms of operator exposure. However, the primary access site for interventional cardiologists has been the right radial artery due to cardiac catheterization laboratories set up for operators to work on the right side of the table. This study seeks to find if a hyperadducted right arm yields less, more, or similar radiation exposure to the operator in cardiac catheterization laboratory than the left radial artery approach.

This study's primary outcome is to measure the radiation exposure to the primary operator during diagnostic cardiac catheterization at four different anatomical locations (these are Maimonides Medical Center employees -attending physicians in the catheterization lab). Study's secondary outcomes aim to measure Dose Area Product, mGy of radiation dose, & contrast administration to the patients undergoing the procedure and presence/absence of subclavian artery tortuosity which are recorded automatically and regardless during the diagnostic procedure.

ELIGIBILITY:
Inclusion Criteria:

* All the Cardiac catheterization laboratory physician operators who consent to participate in the study
* Patients of any sex and gender.
* Age > 18 years old.
* Patients undergoing diagnostic coronary angiogram from in-patient and out-patient settings

Exclusion Criteria:

* History of prior CABG (Coronary Artery Bypass Surgery). CABG patients will be excluded due to inherent increased fluoroscopic time (finding grafts).
* Patients undergoing elective PCI (Percutaneous Coronary Intervention)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: • Patients seen at Maimonides Medical Center, who meet the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Operator radiation exposure | During Cardiac Catheterization
  The primary operators will wear real time radiation dose monitoring at the left eye, right eye, thorax and abdomen level. At the end of each diagnostic procedure the cumulative radiation dose (measured in µSv) data at each level will be collected
Normalized Dose | During Cardiac Catheterization
  The second primary endpoint is Normalized dose, measured by dividing cumulative dose by dose area product (CD/DAP) and entered into query sheet then logged into an Excel spreadsheet.

SECONDARY OUTCOMES:
Dose Area product (DAP) | During Cardiac Catheterization
  Dose area product (DAP) is a quantity used in assessing the radiation risk from diagnostic X-ray examinations and interventional procedures. It is defined as the absorbed dose multiplied by the area irradiated, expressed in gray-centimetres squared.
Flouroscopy time | During Cardiac Catheterization
  Duration of flouroscopy also known as duration of radiation
mGy | During Cardiac Catheterization
  mGy is the unit of absorbed radiation dose
Subclavian tortuosity (Yes/no) | During Cardiac Catheterization
  The anatomic complexity in subclavian artery which causes difficulty in performing cardiac catheterization through radial access.

CONTACTS AND LOCATIONS:
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Pending decision of research committee and any request generated to share data.

REFERENCES:
- [Background] Sciahbasi A, Romagnoli E, Burzotta F, Trani C, Sarandrea A, Summaria F, Pendenza G, Tommasino A, Patrizi R, Mazzari M, Mongiardo R, Lioy E. Transradial approach (left vs right) and procedural times during percutaneous coronary procedures: TALENT study. Am Heart J. 2011 Jan;161(1):172-9. doi: 10.1016/j.ahj.2010.10.003. PMID 21167351
- [Background] Dominici M, Diletti R, Milici C, Bock C, Placanica A, D'Alessandro G, Arrivi A, Italiani M, Buono E, Boschetti E. Operator exposure to x-ray in left and right radial access during percutaneous coronary procedures: OPERA randomised study. Heart. 2013 Apr;99(7):480-4. doi: 10.1136/heartjnl-2012-302895. Epub 2013 Jan 23. PMID 23343690
- [Background] Kado H, Patel AM, Suryadevara S, Zenni MM, Box LC, Angiolillo DJ, Bass TA, Guzman LA. Operator radiation exposure and physical discomfort during a right versus left radial approach for coronary interventions: a randomized evaluation. JACC Cardiovasc Interv. 2014 Jul;7(7):810-6. doi: 10.1016/j.jcin.2013.11.026. Epub 2014 Jun 18. PMID 24954573
- [Background] Sciahbasi A, Frigoli E, Sarandrea A, Calabro P, Rubartelli P, Cortese B, Tomassini F, Zavalloni D, Tebaldi M, Calabria P, Rigattieri S, Zingarelli A, Sardella G, Lupi A, Rothenbuhler M, Heg D, Valgimigli M. Determinants of radiation dose during right transradial access: Insights from the RAD-MATRIX study. Am Heart J. 2018 Feb;196:113-118. doi: 10.1016/j.ahj.2017.10.014. Epub 2017 Oct 28. PMID 29421003
- [Background] Sciahbasi A, Frigoli E, Sarandrea A, Rothenbuhler M, Calabro P, Lupi A, Tomassini F, Cortese B, Rigattieri S, Cerrato E, Zavalloni D, Zingarelli A, Calabria P, Rubartelli P, Sardella G, Tebaldi M, Windecker S, Juni P, Heg D, Valgimigli M. Radiation Exposure and Vascular Access in Acute Coronary Syndromes: The RAD-Matrix Trial. J Am Coll Cardiol. 2017 May 23;69(20):2530-2537. doi: 10.1016/j.jacc.2017.03.018. Epub 2017 Mar 18. PMID 28330794
- [Background] De Rosa S, Torella D, Caiazzo G, Giampa S, Indolfi C. Left radial access for percutaneous coronary procedures: from neglected to performer? A meta-analysis of 14 studies including 7,603 procedures. Int J Cardiol. 2014 Jan 15;171(1):66-72. doi: 10.1016/j.ijcard.2013.11.046. Epub 2013 Nov 23. PMID 24331866
- [Background] Bull JP. Trauma audit. Arch Emerg Med. 1989 Dec;6(4):288-9. doi: 10.1136/emj.6.4.288-b. No abstract available. PMID 2610809
- [Background] Pancholy SB, Joshi P, Shah S, Rao SV, Bertrand OF, Patel TM. Effect of Vascular Access Site Choice on Radiation Exposure During Coronary Angiography: The REVERE Trial (Randomized Evaluation of Vascular Entry Site and Radiation Exposure). JACC Cardiovasc Interv. 2015 Aug 17;8(9):1189-1196. doi: 10.1016/j.jcin.2015.03.026. Epub 2015 Jul 22. PMID 26210808
- [Background] Fu Q, Hu H, Wang D, Chen W, Tan Z, Li Q, Chen B. Randomized comparative study of left versus right radial approach in the setting of primary percutaneous coronary intervention for ST-elevation myocardial infarction. Clin Interv Aging. 2015 Jun 24;10:1003-8. doi: 10.2147/CIA.S81568. eCollection 2015. PMID 26150704
- [Derived] Casazza R, Malik B, Hashmi A, Fogel J, Montagna E, Frankel R, Borgen E, Ayzenberg S, Friedman M, Moskovits N, Verma S, Meng J, Chang N, Huang Y, Rodriguez C, Chera HH, Raj S, Chaterjee S, Gibson D, Palacios A, Agarwal C, Nene MV, Shani J. Operator Radiation Exposure Comparing the Left Radial Artery Approach and a Uniform Hyper-Adducted Right Radial Artery Approach: The HARRA Study. Circ Cardiovasc Interv. 2025 Apr;18(4):e014602. doi: 10.1161/CIRCINTERVENTIONS.124.014602. Epub 2025 Mar 19. PMID 40104858

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT05833516/SAP_000.pdf